CLINICAL TRIAL: NCT01121913
Title: A Randomized, Four-way Crossover Pilot Study to Compare the Relative Bioavailability of Two Prototype Once-a-day Trazodone Hydrochloride Products and Two Marketed Reference Products Following an Equivalent Daily Dose Administration Under Fasting Conditions in Healthy Volunteers
Brief Title: Comparative Bioavailability Study of Two Prototypes of Trazodone Controlled-release Products and Two Marketed Reference Products in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04ACL101
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — Trazodone

ARMS (4):
- Trazodone Contramid® OAD (test product 1) (Experimental): Test product 1 and Test product 2 are two different prototype formulations of Trazodone Contramid® OAD (once a day)
  Interventions: Drug: Trazodone HCl
- Trazodone Contramid® OAD(test product 2) (Experimental): Test product 1 and Test product 2 are two different prototype formulations of Trazodone Contramid® OAD (once a day)
  Interventions: Drug: Trazodone HCl
- Triticco® (Active Comparator)
  Interventions: Drug: Trazodone HCl
- Desyrel® (Active Comparator)
  Interventions: Drug: Trazodone HCl

INTERVENTIONS:
Drug: Trazodone HCl — The dosage of trazodone.HCl during this treatment phase was a single oral dose of 300 mg (one CR tablet) at 07:30 (after an overnight fast of at least 10 hours) on clinic days.
  Arms: Trazodone Contramid® OAD (test product 1)
Drug: Trazodone HCl — The dosage of trazodone.HCl during this treatment phase was a single oral dose of 300 mg (one CR tablet) at 07:30 (after an overnight fast of at least 10 hours) on clinic days.
  Other Names: Oleptro
  Arms: Trazodone Contramid® OAD(test product 2)
Drug: Trazodone HCl — The dosage of trazodone.HCl during this treatment phase was 2 oral doses of 150 mg each: one controlled-release (CR) tablet at 07:30 (after an overnight fast of at least 10 hours) and 19:30 (after a fast of at least 2 hours) on clinic days.
  Arms: Triticco®
Drug: Trazodone HCl — The dosage of trazodone.HCl during this treatment phase was three oral doses of 100 mg each: one immediate-release (IR) tablet at 07:30 (after an overnight fast of at least 10 hours), 15:30 and 23:30 (both dosages after a fast of at least 2 hours) on clinic days.
  Arms: Desyrel®

SUMMARY:
The objectives of this study were:

* to compare the pharmacokinetic profiles of two prototype controlled-release (CR) trazodone hydrochloride (HCl) 300 mg tablets versus two reference products: Trittico® AC (2 x 150 mg CR tablets) and Desyrel® (3 x 100 mg IR (immediate-release) tablets) under fasting condition;
* to assess the controlled release properties of the two prototype formulations;
* to select a prototype formulation for further development;
* to validate the blood sampling schedule for future pivotal pharmacokinetic studies;
* to determine the appropriate sample size for pivotal studies based in the intra-subject variability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18 to 45 years of age (inclusive).
* Body mass within 10% of the ideal mass in relation to height and age, according to the BMI.
* Body mass not less than 70 kg. The normal total circulating blood volume in males and in females is about 71 mL/kg and 65 mL/kg of the body mass, respectively (Meyer, 1988). No subject will have more than 13% of estimated blood volume taken during the study (Standards for the Practice of Blood Transfusion in South Africa, 1999).
* Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the "normal ranges" for the relevant laboratory tests (unless the clinical investigator considers the deviation to be irrelevant for the purpose of the study).
* Normal ECG and vital signs, or abnormalities which the clinical investigator does not consider a disqualification for participation in the study.
* Willingness to undergo pre- and post-study physical examinations, and pre- and post study laboratory investigations.
* Ability to comprehend and willingness to sign both statements of informed consent (for screening and phase-related procedures).
* Non-smoker or past smoker who stopped smoking at least 3 months before entering the study.
* For females, the following conditions are to be met:

  1. has been surgically sterilized, or
  2. is of childbearing potential, and all of the following conditions are met:

     1. had a normal menstrual flow within 1 month before study entry, and
     2. has a negative urine pregnancy test at screening. If this test is positive, the subject will be excluded from the study before receiving study medication. In the rare circumstance that a pregnancy is discovered after the subjects received the study drug, every attempt must be made to follow such subjects to term, and
     3. must agree to use an accepted method of contraception (i.e., spermicide and barrier methods or spermicide and intrauterine contraceptive device). The subject must agree to continue with the same method throughout the study. Hormonal contraceptives will be allowed, with a stable dose for at least one month prior to the first intake of study medication.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* History of, or current compulsive alcohol abuse (> 10 drinks weekly), or regular exposure to other substances of abuse.
* Use of any medication, prescribed or over-the-counter, within 2 weeks prior to the first administration of study medication except if this will not affect the outcome of the study in the opinion of the clinical investigator. Use of hormonal contraceptive agents by females is allowed.
* Participation in another study with an experimental drug within 8 weeks before the first administration of study medication.
* Treatment within the previous 3 months with any drug with a well-defined potential for adversely affecting a major organ or system with evidence to this effect.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity to the study drug or any related drugs.
* History of bronchial asthma.
* History of epilepsy.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of study medication.
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse rate of > 100 beats per minute or < 45 beats per minute during the screening period, either supine or standing.
* Positive testing for HIV, hepatitis B surface antigen and/or Hepatitis C antibodies.
* Positive urine screen for drugs of abuse.
* A urine pregnancy test (ß-HCG) either positive or not performed or lactation.
* Positive urine screen for tobacco use (SureStepTM Smoke Check Tests and One-Step Cotinine (COT) Tests).
* History of marijuana, barbiturate, amphetamine or narcotic abuse within 12 months prior to study start.
* Significant liver disease, defined as active hepatitis or elevated liver enzymes (e.g. aspartate aminotransferase, alanine aminotransferase) >2 times the upper boundary of the normal range.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Primary Completion 2005-04 (Actual)

REFERENCES:
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=17925

RESULTS

PARTICIPANT FLOW:
Groups:
- Trazodone Contramid® OAD (Prototype 1) First: 1 * 300 mg Trazodone Contramid® OAD (prototype 1) tablet test product dosed in treatment phase I; followed by 2 * 150 mg Triticco® tablets (at 07:30 and 19:30) reference product dosed in treatment phase II; 1 * 300 mg Trazodone Contramid® OAD (prototype 2) tablet test product dosed in treatment phase III; and 3 * 100 mg Desyrel® tablets (at 07:30, 15:30 and 23:30) reference product dosed in treatment phase IV. There was a washout period of 7 days between treatment phases.
- Trazodone Contramid® OAD (Prototype 2) First: 1 * 300 mg Trazodone Contramid® OAD (prototype 2) tablet test product dosed in treatment phase I, followed by 1 * 300 mg Trazodone Contramid® OAD (prototype 1) tablet test product dosed in treatment phase II; 3 * 100 mg Desyrel® tablets (at 07:30, 15:30 and 23:30) reference product dosed in treatment phase III; and 2 * 150 mg Triticco® tablets (at 07:30 and 19:30) reference product dosed in treatment phase IV. There was a washout period of 7 days between treatment phases.
- Triticco® First: 2 * 150 mg Triticco® tablets (at 07:30 and 19:30) reference product dosed in treatment phase I; followed by 3 * 100 mg Desyrel® tablets (at 07:30, 15:30 and 23:30) reference product dosed in treatment phase II; 1 * 300 mg Trazodone Contramid® OAD (prototype 1) tablet test product dosed in treatment phase III; and 1 * 300 mg Trazodone Contramid® OAD (prototype 2) tablet test product dosed in treatment phase IV. There was a washout period of 7 days between treatment phases.
- Desyrel® First: 3 * 100 mg Desyrel® tablets (at 07:30, 15:30 and 23:30) reference product dosed in treatment phase I; followed by 1 * 300 mg Trazodone Contramid® OAD (prototype 2) tablet test product dosed in treatment phase II; 2 * 150 mg Triticco® tablets (at 07:30 and 19:30) reference product dosed in treatment phase III; and 1 * 300 mg Trazodone Contramid® OAD (prototype 1) tablet test product dosed in treatment phase IV. There was a washout period of 7 days between treatment phases.
Period: First Intervention Period
Arm/Group | Trazodone Contramid® OAD (Prototype 1) First | Trazodone Contramid® OAD (Prototype 2) First | Triticco® First | Desyrel® First
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: First Washout Period
Arm/Group | Trazodone Contramid® OAD (Prototype 1) First | Trazodone Contramid® OAD (Prototype 2) First | Triticco® First | Desyrel® First
Started | 6 | 6 | 5 | 6
Completed | 5 | 6 | 5 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Trazodone Contramid® OAD (Prototype 1) First | Trazodone Contramid® OAD (Prototype 2) First | Triticco® First | Desyrel® First
Started | 5 | 6 | 5 | 6
Completed | 5 | 6 | 4 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Second Washout Period
Arm/Group | Trazodone Contramid® OAD (Prototype 1) First | Trazodone Contramid® OAD (Prototype 2) First | Triticco® First | Desyrel® First
Started | 5 | 6 | 4 | 6
Completed | 5 | 6 | 3 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Third Intervention Period
Arm/Group | Trazodone Contramid® OAD (Prototype 1) First | Trazodone Contramid® OAD (Prototype 2) First | Triticco® First | Desyrel® First
Started | 5 | 6 | 3 | 6
Completed | 5 | 6 | 3 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Third Washout Period
Arm/Group | Trazodone Contramid® OAD (Prototype 1) First | Trazodone Contramid® OAD (Prototype 2) First | Triticco® First | Desyrel® First
Started | 5 | 6 | 3 | 6
Completed | 4 | 6 | 3 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | Trazodone Contramid® OAD (Prototype 1) First | Trazodone Contramid® OAD (Prototype 2) First | Triticco® First | Desyrel® First
Started | 4 | 6 | 3 | 6
Completed | 4 | 6 | 3 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Trazodone Contramid® OAD (prototype 1) First, Trazodone Contramid® OAD (prototype 2) First, Triticco® First, and Desyrel® First.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Region of Enrollment [Number; unit: participants]
  South Africa | 24

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence Based on AUC(0-t)
Description: AUC(0-t) = Area under the plasma concentration curve vs (versus) time data pairs, where t is the time of the last quantifiable concentration.
  Measured in nanogram x hours per milliliter (ng*h/mL).
Time Frame: 72 hours
Population: The dataset for pharmacokinetic analysis comprised the 19 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Trazodone Contramid® OAD (Prototype 1): 1 * 300 mg Trazodone Contramid® OAD (prototype 1) tablet test product dosed in either treatment phase.
- Trazodone Contramid® OAD (Prototype 2): 1 * 300 mg Trazodone Contramid® OAD (prototype 2) tablet test product dosed in either treatment phase.
- Triticco®: 2 * 150 mg Triticco® tablets (at 07:30 and 19:30) reference product dosed in either treatment phase.
- Desyrel®: 3 * 100 mg Desyrel® tablets (at 07:30, 15:30 and 23:30) reference product dosed in either treatment phase.
Arm/Group | Trazodone Contramid® OAD (Prototype 1) | Trazodone Contramid® OAD (Prototype 2) | Triticco® | Desyrel®
Number analyzed (Participants) | 19 | 19 | 19 | 19
ng*h/mL | 33883 (8069) | 32445 (8868) | 32928 (8313) | 31841 (7398)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD (Prototype 1) vs Triticco®; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LS means) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter AUC(0-t) is between 80% and 125%; Mean ratio = 102, 90% CI 2-sided [91.8 to 114] — Trazodone Contramid® OAD (prototype 1)/Triticco®
Statistical Analysis 2: Comparison: Trazodone Contramid® OAD (Prototype 1) vs Desyrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean ratio = 105, 90% CI 2-sided [93.9 to 117] — Trazodone Contramid® OAD (prototype 1)/Desyrel®
Statistical Analysis 3: Comparison: Trazodone Contramid® OAD (Prototype 2) vs Triticco®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean ratio = 95.3, 90% CI 2-sided [85.5 to 106] — Trazodone Contramid® OAD (prototype 2)/Triticco®
Statistical Analysis 4: Comparison: Trazodone Contramid® OAD (Prototype 2) vs Desyrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean ratio = 97.7, 90% CI 2-sided [87.7 to 109] — Trazodone Contramid® OAD (prototype 2)/Desyrel®

2. Primary Outcome: Bioequivalence Based on AUC(0-∞)
Description: AUC(0-∞) = Area under the plasma concentration curve vs time data pairs, with extrapolation to infinity (∞).
  Measured in nanogram x hours per milliliter (ng*h/mL).
Time Frame: 72 hours
Population: The dataset for pharmacokinetic analysis comprised the 19 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Trazodone Contramid® OAD (Prototype 1) | Trazodone Contramid® OAD (Prototype 2) | Triticco® | Desyrel®
Number analyzed (Participants) | 19 | 19 | 19 | 19
ng*h/mL | 35122 (8655) | 33373 (9299) | 34165 (9105) | 32485 (7621)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD (Prototype 1) vs Triticco®; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LSmeans) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter AUC(0-∞) is between 80% and 125%; Mean ratio = 102, 90% CI 2-sided [91.8 to 114] — Trazodone Contramid® OAD (prototype 1)/Triticco®
Statistical Analysis 2: Comparison: Trazodone Contramid® OAD (Prototype 1) vs Desyrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean ratio = 106, 90% CI 2-sided [95.1 to 118] — Trazodone Contramid® OAD (prototype 1)/Desyrel®
Statistical Analysis 3: Comparison: Trazodone Contramid® OAD (Prototype 2) vs Triticco®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean ratio = 94.9, 90% CI 2-sided [85.1 to 106] — Trazodone Contramid® OAD (prototype 2)/Triticco®
Statistical Analysis 4: Comparison: Trazodone Contramid® OAD (Prototype 2) vs Desyrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean ratio = 98.4, 90% CI 2-sided [88.3 to 110] — Trazodone Contramid® OAD (prototype 2)/Desyrel®

3. Primary Outcome: Bioequivalence Based on Cmax
Description: Cmax = Maximum plasma concentration. Measured in nanogram per milliliter (ng/mL).
Time Frame: 72 hours
Population: The dataset for pharmacokinetic analysis comprised the 19 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Trazodone Contramid® OAD (Prototype 1) | Trazodone Contramid® OAD (Prototype 2) | Triticco® | Desyrel®
Number analyzed (Participants) | 19 | 19 | 19 | 19
ng/mL | 1260 (402) | 1475 (489) | 1688 (442) | 2081 (492)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD (Prototype 1) vs Triticco®; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LSmeans) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter Cmax is between 75% and 133%; Mean ratio = 73.3, 90% CI 2-sided [63.2 to 85] — Trazodone Contramid® OAD (prototype 1)/Triticco®
Statistical Analysis 2: Comparison: Trazodone Contramid® OAD (Prototype 1) vs Desyrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mean ratio = 59.8, 90% CI 2-sided [51.5 to 69.4] — Trazodone Contramid® OAD (prototype 1)/Desyrel®
Statistical Analysis 3: Comparison: Trazodone Contramid® OAD (Prototype 2) vs Triticco®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mean ratio = 83, 90% CI 2-sided [71.5 to 96.4] — Trazodone Contramid® OAD (prototype 2)/Triticco®
Statistical Analysis 4: Comparison: Trazodone Contramid® OAD (Prototype 2) vs Desyrel®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mean ratio = 67.7, 90% CI 2-sided [58.4 to 78.5] — Trazodone Contramid® OAD (prototype 2)/Desyrel®

4. Secondary Outcome: Apparent Terminal Half-life (t½.z)
Description: Apparent terminal half-life (t½.z) of trazodone in hours
Time Frame: 72 hours
Population: The dataset for pharmacokinetic analysis comprised the 19 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Trazodone Contramid® OAD (Prototype 1) | Trazodone Contramid® OAD (Prototype 2) | Triticco® | Desyrel®
Number analyzed (Participants) | 19 | 19 | 19 | 19
Hours | 11.2 (3.92) | 10.9 (3.55) | 10.6 (3.25) | 9.77 (2.49)

5. Secondary Outcome: Time to the Maximum Concentration (Tmax)
Time Frame: 72 hours
Population: The dataset for pharmacokinetic analysis comprised the 19 subjects who completed the study as per protocol.
Measure: Median (Full Range); unit: Hours
Arm/Group | Trazodone Contramid® OAD (Prototype 1) | Trazodone Contramid® OAD (Prototype 2) | Triticco® | Desyrel®
Number analyzed (Participants) | 19 | 19 | 19 | 19
Hours | 12.0 [3.00 to 24.0] | 6.00 [4.00 to 24.0] | 13.0 [2.00 to 16.0] | 8.50 [0.33 to 16.5]

6. Secondary Outcome: Apparent First Order Terminal Rate Constant [λz]
Description: Apparent First order terminal rate constant [λz] of trazodone in plasma expressed in 1/hours.
Time Frame: 72 hours
Population: The dataset for pharmacokinetic analysis comprised the 19 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: 1/hours
Arm/Group | Trazodone Contramid® OAD (Prototype 1) | Trazodone Contramid® OAD (Prototype 2) | Triticco® | Desyrel®
Number analyzed (Participants) | 19 | 19 | 19 | 19
1/hours | 0.07 (0.02) | 0.07 (0.02) | 0.07 (0.02) | 0.08 (0.02)

ADVERSE EVENTS:
Arm/Group | Trazodone Contramid® OAD (Prototype 1) | Trazodone Contramid® OAD (Prototype 2) | Triticco® | Desyrel®
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 7/21 | 9/20 | 14/23 | 14/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trazodone Contramid® OAD (Prototype 1) (N=21) | Trazodone Contramid® OAD (Prototype 2) (N=20) | Triticco® (N=23) | Desyrel® (N=21)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 6 (6) | 6 (7) | 8 (9)
Headache (Nervous system disorders) | 2 (3) | 1 (1) | 4 (5) | 6 (6)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotensive shock (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As reported
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension with convulsions (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — as reported
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The scientific results from this study are the property of the Sponsors, ie, Labopharm Inc., Canada and A.C.R.A.F. S.p.A., Italy. No data reported in the final integrated clinical trial report of this study will be used for publication in scientific journals and/or for presentation at scientific meetings without a previous agreed written consent between the Sponsors.